CLINICAL TRIAL: NCT00367172
Title: Directly Observed Antiretroviral Therapy Among Active Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Frederick L. Altice, MD, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0003011701; R01DA013805 (NIH)
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2009-08

CONDITIONS: HIV/AIDS; Substance Abuse
Keywords: human immunodeficiency virus; acquired immunodeficiency syndrome; substance abuse; directly administered antiretroviral therapy; adherence, directly observed therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Directly Observed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Directly Administered Antiretroviral Therapy

SUMMARY:
The goal of this randomized, controlled trial is to compare the effectiveness of a community-based program of providing supervised antiretroviral therapy to HIV-positive drug users, compared to having the patients take the medicines on their own.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has dramatically reduced morbidity and mortality from HIV disease, but these benefits have not been conferred equally among all patient populations. Injection drug users (IDUs) have shown particularly less favorable outcomes, with HIV progression remaining at high levels, and IDU remains a significant risk behavior for the spread of HIV worldwide, with explosive epidemics in Eastern Europe, Russia, and Southeast Asia. It is therefore essential to develop and test strategies of HIV treatment that optimize outcomes for this population, in order to reduce morbidity and mortality and to curb secondary transmission.

Directly observed therapy (DOT) for tuberculosis has resulted in impressive improvements in adherence and clinical response and marked reductions in the development of resistance. The time-limited treatment of tuberculosis, the inherently different transmission patterns of tuberculosis and HIV, and the complexity of antiretroviral therapy have raised concerns about translating the DOT model to HIV. Successful, but non-comparative demonstration programs of directly administered antiretroviral therapy (DAART) have been implemented in methadone maintenance programs, community-based settings, skilled nursing facilities, and in prisons. None of these, however, have targeted active drug users or used a prospective, randomized controlled trial (RCT) design to rigorously determine the efficacy of DAART as an intervention to improve HIV outcomes among active drug users. One RCT of DAART recently failed to demonstrate an impact on virological outcomes among low-income HIV+ patients, but these results are unlikely to be applicable to IDUs or other populations with demonstrated problematic adherence.

We therefore conducted the first randomized controlled trial to address this question, consisting of six months of DAART versus self-administered therapy (SAT) among active drug users in a community setting. The objective was to determine the potential efficacy of a six-month DAART program on HIV infection, using surrogate markers of HIV- RNA levels and CD4+ T lymphocyte counts.

ELIGIBILITY:
Inclusion Criteria:

1. being HIV seropositive;
2. being eligible for and/or being prescribed HAART
3. living within the city of New Haven
4. actively using heroin and/or cocaine in the previous six months
5. receiving no more than a twice-daily regimen

Exclusion Criteria:

Not meeting inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2001-06; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Virological Success, defined as greater than 1 Log HIV-1 Copies/mL reduction or Viral Load Less than 400 copies/mL at the end of six months on the intervention.

SECONDARY OUTCOMES:
Mean change in HIV-1 viral load from baseline to six months at the end of the intervention.
Virological Success at six months following the termination of the intervention.
3-Day Recall measures of adherence at the end of six months on the intervention.
Mean change in HIV-1 viral load from baseline six months following the termination of the intervention.
Mean change in CD4+ T cells from baseline to the end of six months on the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, M.D., Principal Investigator — Yale AIDS Program; Gerald H Friedland, Principal Investigator — Yale AIDS Program
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Altice FL, Mezger JA, Hodges J, Bruce RD, Marinovich A, Walton M, Springer SA, Friedland GH. Developing a directly administered antiretroviral therapy intervention for HIV-infected drug users: implications for program replication. Clin Infect Dis. 2004 Jun 1;38 Suppl 5:S376-87. doi: 10.1086/421400. PMID 15156426
- [Derived] Altice FL, Maru DS, Bruce RD, Springer SA, Friedland GH. Superiority of directly administered antiretroviral therapy over self-administered therapy among HIV-infected drug users: a prospective, randomized, controlled trial. Clin Infect Dis. 2007 Sep 15;45(6):770-8. doi: 10.1086/521166. Epub 2007 Aug 13. PMID 17712763